CLINICAL TRIAL: NCT04937608
Title: Impact of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection on the Sperm Parameters of Infertile Men
Brief Title: Impact of the Coronavirus Disease 2019 (COVID-19) on Sperm Parameters
Status: Terminated | Type: Observational
Why Stopped: Lack of staff
Sponsor: Fertilys (Industry)
Collaborators: Institut national de la recherche scientifique (Unknown)
Responsible Party: Sponsor
Other Study IDs: COVID-19 and sperm parameters
Record Dates: First submitted 2021-06-21; First posted 2021-06-24 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Covid19; Infertility, Male
MeSH Terms: conditions — COVID-19; Infertility, Male

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 group: men aged 18 to 45 who have been infected with SARS-CoV-2 in the past 6 months
  Interventions: Diagnostic Test: Sperm analysis
- Control group: healthy men aged 18 to 45 with normal sperm parameters (WHO 2010 criteria) and who have never contracted COVID-19
  Interventions: Diagnostic Test: Sperm analysis

INTERVENTIONS:
Diagnostic Test: Sperm analysis — Routine sperm analysis including analysis of sperm concentration, motility, vitality and morphology. Sperm DNA integrity will also be assessed.

SUMMARY:
This study aims to better understand the effects of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, virus that causes the coronavirus disease 2019 (COVID-19), on male fertility.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will produce a sperm sample by masturbation. Patients will also complete a questionnaire relating to their state of health. Six month following the first sperm sample, patients will produce another sperm sample by masturbation. These sperm parameters will be compared with the ones from a sperm analysis performed less than 2 years before the SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* All men aged 18 to 45 having a sperm analysis done at the Fertilys fertility center in the last 2 years who have not contracted COVID-19, agreeing to participate in the study and having signed the consent form to participate in the study.
* All men aged 18 to 45 having a sperm analysis done at the Fertilys fertility center in the last 2 years) who have contracted COVID-19 within the last 6 months, agreeing to participating in the study and having signed the consent form to participate in the study.
* All men aged 18 to 45 years with a sperm concentration ≥ 15 million/mL, progressive motility ≥ 20% and a percentage of normal forms ≥ 2%.

Exclusion Criteria:

* Men aged under 18 and over 45.
* Men who cannot produce a sperm sample by antegrade ejaculation.
* Men whose sperm concentration is <15 million/mL, progressive motility <20% and a percentage of normal forms <2%, determined following the production of a "reference" sperm sample, carried out before March 2020, i.e. before the COVID-19 pandemic.

Ages: 18 Years to 45 Years | Sex: Male
Age Groups: Adult
Study Population: See Eligibility Criteria
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in sperm parameters quality | Pre-infection, on the day of recruitment and six month later
  Sperm concentration and motility will be assessed using computer-assisted sperm analysis (CASA). Sperm vitality and morphology will be evaluated using eosine-nigrosine and Romanowsky staining techniques, respectively. DNA fragmentation and sperm chromatin decondensation will be measured using the Terminal deoxynucleotidyl transferase dUTP nick end labeling (TUNEL) and aniline blue assays, respectively. These sperm parameters will be compared before and after SARS-CoV-2 infection and between the different time frames.
Viral RNA in seminal plasma | Pre-infection, on the day of recruitment and six month later
  The number of SARS-CoV-2 RNA copies and viral particles / mL of seminal plasma will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Fertilys, Laval, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No